CLINICAL TRIAL: NCT01854801
Title: Evaluation of a Specialized Therapeutic Care of Patients Presenting an Idiopathic Environmental Intolerance Attributed to Electromagnetic Fields
Brief Title: Evaluation of a Specialized Therapeutic Care of Patients Presenting an Intolerance Attributed to Electromagnetic Fields
Acronym: IEI-CEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANSES, France (Unknown); INERIS, Verneuil-En-Halatte, France (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100120
Record Dates: First submitted 2013-04-24; First posted 2013-05-16 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Environmental Intolerance Attributed to Electromagnetic Fields
Keywords: IEI-EMF; WI-FI; DECT; Electro-sensitivity; Radiofrequency; EHS; Idiopathic; Environmental; Intolerance fields; Mobile phone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Patients who declare themselves to be intolerant to electromagnetic fields benefit from medical care in occupational and environmental diseases centers and from a measurement of individual electromagnetic exposures and symptoms episodes. Each patient is his own control.
  Interventions: Other: Individual medical Care; Other: Individual electromagnetic exposures

INTERVENTIONS:
Other: Individual medical Care — Individual medical care in occupational and environmental diseases centers
Other: Individual electromagnetic exposures — During 7 days, patient hold a dosimeter measuring their electromagnetic exposures for FM, TV, GSM, DECT, WIFI, TETRA and relay antenna emissions. During this week, patients notify intensity and time of their symptoms on a self-questionary

SUMMARY:
The purpose of the study is to evaluate efficacy of a 14 months follow-up and individual medical care of electro-sensitive patients: by measurement of health status, sensitivity to electromagnetic fields exposures, and quality of life.

DETAILED DESCRIPTION:
110 patients suffering from Idiopathic Environmental Intolerance attributed to electromagnetic fields (IEI-EMF) are expected in this trial.

Type of trial: Interventional multicenter study, non-randomized, with measurement before and after intervention. Each patient is his own control.

Primary outcome: Efficacy of an individual medical care on electro sensitive (IEI CEM) patients evaluated from the improvement of health status, sensitivity to electromagnetic fields (EMF) exposure, and quality of life.

Scheme:

Visit 1(T0): Patients undergo a specialized medical examination: a standardized medical record is filled in. Physicians evaluate the psychological impact of IEI-EMF and a psychotherapeutic care is proposed if necessary. Patients fill in 2 self-questionaries: quality of life (SF-36) and EMF exposure sensitivity.

After the visit 1, a symptoms self-administrated questionary n°1 is completed during 7 days.

1 month after inclusions (T1), radiofrequencies (RF) are recorded by a dosimeter worn by patients for 7 days; patient fill-in the symptoms self-administrated questionary n° 2 during the same time.

Visit 2: 6 months after inclusion, analysis of symptoms and RF exposure is restituted at patient. An adapted care is proposed.

12 months after inclusion (T12), patients complete the symptoms self-administrated questionary n°3.

Visit 3: 14 months after inclusion (T14), patients have medical examination and complete the quality of life and EMF exposure sensitivity self-questionaries. Standardized medical record is filled in by physicians. Patient and physician discuss the global and comparative analysis of individual results.

Inclusion duration: 24 month; Follow-up: 14 months; Study duration: 38 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who declare themselves to be intolerant to electromagnetic fields
* Subjects over 18 years old
* Subjects affiliated to a social security scheme
* Subjects who signed the consent form

Exclusion Criteria:

* Subject with a disorder of the understanding of the French language at the discretion of the investigator
* Pregnant women,
* Persons deprived of their liberty, persons under guardianship, and persons in emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-03-09 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Measurement of symptoms severity | At 12 months after inclusion .
  At month 12 months the severity of symptoms is evaluated by a self-questionary filled in during 7 days. The level of severity of each symptom occurring during a week, will be self-evaluated by the patient on the base of a 0 to 5 scale. Following the intervention we expect a reduction in the severity of symptoms described.
Measurement of symptoms frequency | At 12 months after inclusion
  At month 12 months the symptoms frequency is evaluated by a self-questionary filled in during 7 days. Each symptom occurring during a week is reported by the patient allowing calculation of a frequency in symptoms appearance. Following the intervention we expect a reduction in the frequency of symptoms described.
Sensitivity to electromagnetic fields | at 14 months
  At visit 3 (14 months) the EMF sensitivity is evaluated by the self-questionary.
Measurement of symptoms frequency | At 1 month after inclusion
  At month 1 months the symptoms frequency is evaluated by a self-questionary filled in during 7 days. Each symptom occurring during a week is reported by the patient allowing calculation of a frequency in symptoms appearance. Following the intervention we expect a reduction in the frequency of symptoms described.
Measurement of symptoms severity | At 1 month after inclusion
  At month 1 month the severity of symptoms is evaluated by a self-questionary filled in during 7 days. The level of severity of each symptom occurring during a week, will be self-evaluated by the patient on the base of a 0 to 5 scale. Following the intervention we expect a reduction in the severity of symptoms described.
Sensitivity to electromagnetic fields | at day 0
  At visit 1 (day 0), the EMF sensitivity is evaluated by the self-questionary.

SECONDARY OUTCOMES:
Quality of life evaluation | at 14 months.
  At visit 3 (14 months), the quality of life is evaluated by the self-questionary (SF-36)
Compliance to the study design | At each Visit (Day 0, Month 1, Month 6 and month 14)
Quality of life evaluation | day 0
  At visit1 (day 0), the quality of life is evaluated by the self-questionary (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda BENSEFA-COLAS, MD, Study Director — Service de Pathologie Professionnelle, Hopital Cochin, AP-HP, Paris; Rene de SEZE, MD, Study Director — INERIS (Institut National de l'EnviRonnement Industriel et des RisqueS)
Locations (1):
- Service de Pathologie Professionnelle, Hôpital Cochin, Hôpitaux Universitaires Paris Centre, Paris, France

REFERENCES:
- See also: The link presents the recruiting centers — http://www.radiofrequences.gouv.fr/spip.php?article102